CLINICAL TRIAL: NCT05256680
Title: The Effect of Gardening Activities Applied to The Elderly in Nursing Home on Psychological Wellness and Depression: A Single Blind Randomized Controlled Study
Brief Title: Gardening Activities for the Elderly Psychological Well-Being and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Head of Public Health Nursing Department, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ordu1234
Record Dates: First submitted 2022-02-03; First posted 2022-02-25 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Elderly Person

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gardening Activities (Experimental): In the research, the elderly in the experimental group will have gardening activities once a week for 3 months.
  Interventions: Other: Gardening Activities
- Control (Active Comparator): No intervention will be applied to the elderly in the control group during the research. They will participate in routine activities in the nursing home.
  Interventions: Other: Gardening Activities

INTERVENTIONS:
Other: Gardening Activities — In the research, the elderly in the experimental group will have gardening activities once a week for 3 months.
  No intervention will be applied to the elderly in the control group during the research. They will participate in routine activities in the nursing home.

SUMMARY:
Purpose of the Study: This research will be conducted to determine the effects of gardening activities applied to the elderly in nursing homes on psychological well-being and depression.

Research Hypotheses H0: Gardening activities applied to the elderly in the nursing home do not affect the psychological well-being of the elderly.

H1: Gardening activities applied to the elderly in nursing homes increase the psychological well-being of the elderly.

H0: Gardening activities applied to the elderly in the nursing home do not affect the depression level of the elderly.

H1: Gardening activities applied to the elderly in nursing homes reduce the depression level of the elderly.

DETAILED DESCRIPTION:
This study was planned as a single-blind randomized controlled experimental study.

ELIGIBILITY:
Inclusion Criteria:

* Staying in a nursing home for at least 3 months,
* Does not have a physical disability that may hinder gardening activities,
* No vision or hearing loss that may hinder gardening activities,
* Open to communication and cooperation,
* The elderly who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Having a serious medical disability (such as paralysis, Parkinson's),
* Having a serious psychiatric diagnosis,
* Severely demented and
* The elderly who do not want to continue the research will be excluded from the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Psychological Well-Being Scale | 12 weeks
  The Turkish validity and reliability studies of the scale, which was developed by Butler and Kern (2016), in order to evaluate the well-being levels of individuals, were conducted by Demirci et al. (2017), made by The scale consists of 15 items, 8 fillers and 5 sub-dimensions.
  In the evaluation of the scale, the average score of the items of each dimension is taken. However, none alone explains the level of well-being; each dimension contributes to well-being. In addition, apart from the dimensions of well-being, Butler and Kern (2016) stated that 6 of the 8 fillers in the scale were H health (4th, 13th and 18th items) and N negative emotions (7th, 14th and 20th items). added as a separate size.
Geriatric Depression Scale | 12 weeks
  Yesavage et al. (1993) based on self-report. The short form of GDS consisting of 15 questions will be used in this study. The Turkish validity and reliability study of the scale was performed by Ertan et al. (1997), by 5 questions (1st, 5th, 7th, 11th and 13th) in the scale are structured positively and the others negatively. In the evaluation of the scale, "no" answers to positive questions and "yes" answers to negative questions were matched with 1 point each. The scores that can be obtained from the scale are between 0-15. Above five points is considered as depression. The cronbach alpha value of the scale is 0.92.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GÖK UĞUR, Assoc. Dr., Principal Investigator — Ordu University; Şeyma ŞENGÜR, PhD, Study Director — Ordu University
Locations (1):
- Hacer GOK UGUR, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No